CLINICAL TRIAL: NCT03988777
Title: Magnetic Seed Localisation for Nonpalpable Breast Lesions: a Combined Retrospective and Prospective Analysis
Brief Title: Magnetic Seed Localisation for Nonpalpable Breast Lesions
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S61864
Record Dates: First submitted 2019-05-29; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-05

CONDITIONS: Oncology; Breast Cancer
Keywords: Breast cancer; Nonpalpable breast lesions; Hooked-wire localisation; Magnetic seed localisation
MeSH Terms: conditions — Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Prospective Magseed: This cohort includes patients with an impalpable breast lesion that are scheduled for breast conserving surgery with Magseed localisation after September 2018. Their data will be prospectively collected and analysed.
  Interventions: Device: Preoperative localisation technique
- Retrospective hooked-wire: This cohort includes patients with an impalpable breast lesion that were scheduled for breast conserving surgery with hooked-wire before September 2018. Their data will be retrospectively collected and analysed.
  Interventions: Device: Preoperative localisation technique

INTERVENTIONS:
Device: Preoperative localisation technique — Impalpable breast lesions are preoperatively localised, either with hooked-wire (retrospective study) or Magseed (prospective study)

SUMMARY:
Screening programs and advances in imaging have led to more breast lesions being diagnosed at an impalpable stage. Multiple localisation techniques for nonpalpable breast lesions have been developed during the past decades. Specifically, several alternatives to the golden standard hooked-wire technique have become available, of which magnetic seed localisation is one of the newest approaches. Since September 2018, Magseed® localisation is the standard of care for localising impalpable breast lesions in UZ Leuven. In this study, the oncological safety, the clinical safety and surgeon satisfaction of Magseed® localisation will be assessed and retrospectively compared to hooked-wire localisation.

ELIGIBILITY:
Inclusion Criteria:

* Breast conserving surgery with preoperative localisation
* Minimum 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population includes women (18+) with an impalpable breast lesion suitable for breast conserving surgery.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Number of participant with device-related adverse events | Up to three weeks after surgical treatment
Total breast volume resected during breast conserving surgery | Up to three weeks after surgical treatment
Number of participants with positive surgical margins as assessed by pathological examination of the specimen | Up to three weeks after surgical treatment
Re-operation rate due to positive surgical margins | Up to three weeks after surgical treatment
Surgeon satisfaction based on a questionnaire | After surgery
  After surgery, the surgeon will be asked to describe the magnetic seed procedure, choosing between 'easier than hooked-wire' or 'more challenging than hooked-wire'. Moreover, the surgeon wil have the chance to add additional remarks or experiences with this new technique.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No